CLINICAL TRIAL: NCT01776762
Title: Effect of Nutritional Intervention in a Cross-sector Model for the Rehabilitation of Undernourished Geriatric Medical Patients: a Randomized Controlled Trial.
Brief Title: Nutritional Intervention in a Cross-sector Model for the Rehabilitation of Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christian Bitz, Head of research, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFFECT.B01.2012
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Malnutrition
Keywords: Nutrition; Rehabilitation; Weightloss
MeSH Terms: conditions — Malnutrition; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual nutritional therapy (Experimental): Individual nutritional therapy provided by registered dietician by means of three Home-visits
  Interventions: Dietary Supplement: Individual nutritional therapy
- Standard Follow-home programme (No Intervention): Standard Follow-home programme without individual nutritional therapy

INTERVENTIONS:
Dietary Supplement: Individual nutritional therapy — Individual nutritional therapy provided by registered dietician by means of three Home-visits
  Arms: Individual nutritional therapy

SUMMARY:
Based on an established Follow-home-programme offered at discharge from hospital the aim of this study is to test a model of how nutritional intervention in elderly patients can be systematized and quality assured in the transition between sectors. Furthermore the aim is to demonstrate that this model has a positive effect on the functioning and well-being of the elderly patient.

The purpose of the Follow-home-programme is to facilitate the transition of the elderly patient between hospital and private home in order to follow-up on any medical, nursing- or retraining-related intervention necessary to the rehabilitation of the patient. However this offer does not focus on nutrition in particular. This is a problem as many elderly patients are known to develop a poor nutritional status due to low appetite, disease etc. Our hypothesis is that adding a systematic nutritional focus to the Follow-home intervention programme will promote the rehabilitation of the elderly patient further.

The nutritional intervention in our study will focus on improving energy- and protein intake and we will measure the effect on the patient's functional abilities, quality of life and rate of hospital readmissions. The intervention model will be based on individualized nutritional counselling by a registered dietician in the patients home.

DETAILED DESCRIPTION:
The study is designed as a 12 week randomized, controlled intervention study. The study sample will consist of 80 geriatric patients admitted to a medical ward at Herlev University Hospital in Copenhagen, Denmark. The patients will be equally distributed into the control and the intervention group. The control group will follow the usual follow-home programme. The intervention group will also follow this programme, but will additionally be offered 3 home visits by a registered dietician. Interdisciplinary information exchange will take place through established communication channels eg. patient records, visitations.

Before and after the intervention data on the patient eg. hand-grip strength, nutritional status, dietary intake, functional abilities, well-being and activities of daily living will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric medical patients
* Age +70 years
* Nutritional risk according to the level 1 screen in Nutritional Risk Screening 2002 (NRS2002)
* Nutritional therapy for at least 3 days and at least in two daily meals during the hospitalization period
* Participation in the standard Follow-home programme

Exclusion Criteria:

* Dementia
* Expected readmissions
* Terminal disease
* Non-danish speaking
* Not able to perform Hand grip test
* Planning weight reducing diet

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 12 weeks

SECONDARY OUTCOMES:
Functional status | 12 week
  Chair stand, mobility, disability and rehabilitation capacity
Nutritional status | 12 weeks
  Weight, BMI, energy and protein intake, distribution of protein intake
Need of social services | 12 weeks
  Home care, home nursing, meals-on-wheels
Readmissions | 6 months before and 1½ year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christian Bitz, Cand Scient, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- EFFECT, Copenhagen University Hospital at Herlev, Herlev, Copenhagen, Denmark

REFERENCES:
- [Background] Beck A, Rask KØ, Leedo E, Jensen LL, Martins K, Vedelspang A (2014) Study Protocol: Nutritional Support in a Cross-sector Model for the Rehabilitation of Geriatric Patients: A Randomized Controlled Trial. J Clin Trials 4: 165.
- [Background] Pohju A, Belqaid K, Brandt C, Lugnet K, Nielsen AL, et al. (2016) Adding a Dietitian to a Danish Liaison-Team after discharge of geriatric patients at nutritional risk may save health care costs. Aging Sci 4: 159.
- [Result] Beck A, Andersen UT, Leedo E, Jensen LL, Martins K, Quvang M, Rask KO, Vedelspang A, Ronholt F. Does adding a dietician to the liaison team after discharge of geriatric patients improve nutritional outcome: a randomised controlled trial. Clin Rehabil. 2015 Nov;29(11):1117-28. doi: 10.1177/0269215514564700. Epub 2014 Dec 31. PMID 25552522